CLINICAL TRIAL: NCT00814788
Title: Phase II Trial of Bicalutamide and RAD001 in Patients With Hormone-Independent Prostatic Adenocarcinoma (HIPC) After the First-Line Androgen Deprivation Therapy
Brief Title: Bicalutamide With or Without Everolimus in Treating Patients With Recurrent or Metastatic Prostate Cancer
Acronym: UCDCC#215
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCDCC#215; 223646 (Other Grant/Funding Number: UC Davis); Novartis (Other Grant/Funding Number: CRAD001CUS53T)
Record Dates: First submitted 2008-12-24; First posted 2008-12-25 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Prostate Cancer
Keywords: stage IV prostate cancer; adenocarcinoma of the prostate; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bicalutamide + Everolimus (Experimental): Patients receive oral bicalutamide and oral everolimus once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bicalutamide; Drug: Everolimus

INTERVENTIONS:
Drug: Bicalutamide — 50 mg oral tablet daily
  Other Names: Casodex
Drug: Everolimus — 10 mg oral capsule daily
  Other Names: Afinitor; RAD001

SUMMARY:
RATIONALE: Androgens can cause the growth of prostate cancer cells. Antihormone therapy, such as bicalutamide, may lessen the amount of androgens made by the body. Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying bicalutamide and everolimus to see how well they work compared with bicalutamide in treating patients with recurrent or metastatic prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To compare the PSA response rate in patients with hormone-independent recurrent or metastatic adenocarcinoma of the prostate treated with bicalutamide and everolimus after first-line androgen deprivation therapy.
* To evaluate the time to treatment failure and overall survival of these patients.
* To assess the toxicity of bicalutamide and everolimus in these patients.

OUTLINE: Patients are stratified according to disease status (metastatic disease vs biochemical recurrence without measurable disease).

Patients receive oral bicalutamide and oral everolimus once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 28-42 days and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria

1. Participants must be adult males >18 years.
2. Patients must have histologically or cytologically confirmed CaP with a Gleason score available or interpretable.
3. Patients must have CaP deemed to be androgen independent.
4. Measurable disease is not required.
5. Patients must have been surgically or medically castrated. If the method of castration was LHRH agonists (leuprolide or goserelin) or antagonists (degarelix), then the patient must be willing to continue the use of LHRH agonists or antagonists. Serum testosterone must be at castrate levels (< 50 ng/dL) within 3 months prior to registration.
6. Participant has not been on any previous therapy with androgen receptor antagonists or mTOR inhibitors. Note: patients who have taken an androgen receptor antagonist for a brief period (no more than 2 months) at the start of LHRH agonist therapy to prevent flare will be considered eligible.
7. Men enrolled in this trial must agree to use adequate contraception prior to study entry and for the duration of study participation.
8. Patients must have normal organ and marrow function.
9. Ability to understand and the willingness to sign a written informed consent document
10. ECOG performance status 0-2.
11. Patients having any respiratory symptoms such as cough and shortness of breath have undergone pulmonary function testing revealing no worse than mild impairment.

Exclusion Criteria

1. No documented histological confirmation of CaP.
2. Patient has received other hormonal therapy besides first-line androgen deprivation therapy with LHRH agonist, LHRH antagonist, orchiectomy, high-dose steroid, abiraterone, provenge and ketoconazole.
3. Patients who have received prior treatment with an mTOR inhibitor.
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
5. HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with RAD001.
6. Patients currently receiving anticancer therapies or who have received anticancer therapies within 4 weeks of the start of study drug (including chemotherapy, radiation therapy, antibody based therapy, etc.)
7. Patients who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia) or patients that may require major surgery during the course of the study.
8. Prior treatment with any investigational drug within the preceding 4 weeks.
9. Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent.
10. Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period.
11. Patients on herbs or other alternative medicines for the treatment of prostate cancer, including but not limited to saw palmetto, PC-SPES.
12. Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases.
13. Other malignancies within the past 3 years except for adequately treated basal or squamous cell carcinomas of the skin or other Stage 0 or I cancers.
14. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001.
15. Patients with an active, bleeding diathesis.
16. History of noncompliance to medical regimens.
17. Patients unwilling to or unable to comply with the protocol.
18. Patients with active pulmonary disorders or history of moderately to severely impaired pulmonary function tests will be excluded from the study.
19. Patients with symptomatic metastatic prostate cancer such as moderate to severe pain, impaired organ function or spinal cord compression will be excluded from this study unless these issues have been taken care of.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-12; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chong-Xian Pan, MD, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Cancer Center, Sacramento, California, United States

REFERENCES:
- [Background] Chow H, Ghosh PM, deVere White R, Evans CP, Dall'Era MA, Yap SA, Li Y, Beckett LA, Lara PN Jr, Pan CX. A phase 2 clinical trial of everolimus plus bicalutamide for castration-resistant prostate cancer. Cancer. 2016 Jun 15;122(12):1897-904. doi: 10.1002/cncr.29927. Epub 2016 Mar 28. PMID 27019001

RESULTS

PARTICIPANT FLOW:
Groups:
- Bicalutamide + Everolimus: Patients receive oral bicalutamide and oral everolimus once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Bicalutamide 50 mg oral daily
  Everolimus: RAD001 10 mg oral capsule daily - continuously.
Period: Overall Study
Arm/Group | Bicalutamide + Everolimus
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Bicalutamide + Everolimus: Patients receive oral bicalutamide and oral everolimus once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  bicalutamide: Bicalutamide 50 mg oral daily
  Everolimus: RAD001 10 mg oral capsule daily - continuously.
Arm/Group | Bicalutamide + Everolimus
Number analyzed (Participants) | 24
Age, Continuous [Mean (Full Range); unit: years] | 71.1 [53 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 24
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: PSA Response Rate
Description: The PSA response rate was defined as a 30% reduction in the PSA level from baseline. PSA Working Group consensus criteria combined with radiographic studies were used to determine the proportion of patients with PSA decline.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Bicalutamide + Everolimus
Number analyzed (Participants) | 24
Participants | 18

2. Secondary Outcome: Progression-free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bicalutamide + Everolimus
Number analyzed (Participants) | 24
months | 9.4 [4 to 25]

3. Secondary Outcome: Overall Survival
Description: Overall survival was estimated using the Kaplan-Meier method.
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bicalutamide + Everolimus
Number analyzed (Participants) | 24
months | 28 [14.1 to 42.7]

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Bicalutamide + Everolimus
All-Cause Mortality (participants affected / at risk) | 2/24
Serious Adverse Events (participants affected / at risk) | 1/24
Other Adverse Events (participants affected / at risk) | 17/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bicalutamide + Everolimus (N=24)
Sepsis (General disorders) | 1 (1) — Nonneutropenic sepsis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bicalutamide + Everolimus (N=24)
Anemia (Blood and lymphatic system disorders) | 14 (14)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
ALT increase (Hepatobiliary disorders) | 4 (4)
ALK phosphastase increased (Hepatobiliary disorders) | 6 (6)
Anal mucositis (General disorders) | 1 (1)
Anorexia (Psychiatric disorders) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
AST increased (Hepatobiliary disorders) | 8 (8)
Constipation (Gastrointestinal disorders) | 3 (3)
Constitutional Symptoms (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Dry mouth (General disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Deep Vein Thrombosis (Vascular disorders) | 1 (1)
Edema (Blood and lymphatic system disorders) | 6 (6)
Fatigue (General disorders) | 16 (16)
Hand Foot Syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Hypercholesterolemia (Cardiac disorders) | 15 (15)
Hyperglycemia (Renal and urinary disorders) | 12 (12)
Hypertriglyceridemia (Cardiac disorders) | 13 (13)
Leukopenia (Blood and lymphatic system disorders) | 17 (17)
Lymphopenia (Blood and lymphatic system disorders) | 16 (16)
Oral mucositis (Skin and subcutaneous tissue disorders) | 14 (14)
Neutropenia (Blood and lymphatic system disorders) | 9 (9)
Nausea (Gastrointestinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Proteinuria (Blood and lymphatic system disorders) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 5 (5)
Right hip pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 2 (2)
Taste Alteration (General disorders) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (8)
Weight Loss (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes